CLINICAL TRIAL: NCT00519922
Title: Efficacy of Kinesthesia, Balance and Agility Exercise Training as Treatment of Knee Osteoarthritis: A Pilot Study
Brief Title: A Study of the Effectiveness of Different Types of Exercise for People With Knee Osteoarthritis
Acronym: KBA Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Arthritis Research Institute of America (Other)
Responsible Party: Matthew W Rogers, Director of Exercise Research, The Arthritis Research Institute of America
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KneeOAExercise-1
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Kinesthesis; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): KBA = Kinesthesia, Balance, Agility Exercise Training
  Interventions: Other: Kinesthesia, Balance, and Agility (KBA) Exercise
- 2 (Active Comparator): Standard Lower Extremity Strength Training
  Interventions: Other: Standard LE Strength Training

INTERVENTIONS:
Other: Kinesthesia, Balance, and Agility (KBA) Exercise — Participants will exercise three times per week 20 to 30 minutes per session. Agility/Active Range of Motion exercises provide warm-up, improve joint range-of-motion & agility, dynamic proprioception,functional strength & endurance.
  Kinesthesia & Balance Training will challenge the subject's proprioceptive and neuromuscular control mechanisms to adapt and stabilize the knee joints during dynamic ADL activities (walking, climbing, etc); improve static and dynamic balance and sense of stability & confidence in ADL activities.
  Soft pads will be used to progress some of the kinesthesia & balance challenge training. Thera-Band® balance pads at 3 levels of softness will be used. These balance pads allow both appropriate starting difficulty and progression of difficulty level (i.e., the softer the pad, the greater the difficulty). Subjects will demonstrate safe balance on a stable surface (i.e. one-footed standing on floor) prior to progressing to the first level of the soft pads.
  Arms: 1
Other: Standard LE Strength Training — Standard therapeutic exercises for knee OA which are widely used. Body weight and Thera-Band® color coded elastic bands will be used as appropriate to provide resistance. Exercises will be progressed according to the individual participant's improvement. All training for the ST condition will be conducted on stable surfaces (e.g. standing on floor, sitting in chair, lying on floor). Exercises may include 4-direction straight leg lifts, heel slides, quad sets, internal & external hip rotation, heel raises, toe raises, knee extension, knee flexion, partial squats/wall slides, etc.
  Arms: 2

SUMMARY:
This pilot study will test the testing and exercise training protocols for a larger study that is in the desing phase and may be modified based on the findings of this study. Two exercise groups will be compared; one is a stadard treatment group using leg strength exercises that are commonly employed in therapy clinics. The other group will do balance and agility type exercises, but no specific strength exercises. These "KBA" exercises are increasingly common in therapy clinics, but very little research has been conducted on their effectiveness in treating knee osteoarthritis symptoms. Participants in this study will complete three short paper and pencil tests at the beginning and end of the study (8 weeks of exercise) as well as a leg strength test, a leg endurance test, two short walking tests, and a stair climb/descend test. One of the paper and pencil tests will be taken every two weeks in an effort to see how quickly changes to symptoms might occur. The exercise programs will be conducted 3 afternoons per week (Mon-Wed-Fri) and will be lead by an ACSM certified instructor.

DETAILED DESCRIPTION:
Radiographic knee OA is present in an estimated 37% of Americans over the age of 60, representing more than 13 million people. Current medical, non-surgical knee OA treatments focus primarily on symptomatic relief and have met with limited, temporary success. Various therapeutic exercise prescriptions have been used to help ameliorate knee OA symptoms and improve function. Leg strength training is most commonly used. However, recent evidence suggests that shorter programs of kinesthesia, balance and agility (KBA) techniques may result in more rapid symptom relief and functional improvements in comparison to traditional therapeutic exercise. These early benefits could potentially lead to greater long term exercise adherence.

In a case study of an elderly female patient with dynamic knee instability related to OA, physical therapists reported success with a combination of KBA training and traditional therapeutic exercise. These findings need to be verified in a controlled clinical trial. This pilot study will help determine the proper testing and exercise training methods for a larger clinical trial, and will indicate if KBA training done without concurrent strength training is a viable intervention.

Research Hypothesis: Among men and women age 50 and over with Kellgren and Lawrence (1957) Grade 2 or higher symptomatic tibiofemoral OA in one or both knees, an 8-week, 3-day per week kinesthesia, balance & agility (KBA) exercise program - designed to increase dynamic neuromuscular knee stability - safely and effectively changes physical function more effectively than standard leg strength training

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or over of either gender
* Radiographic tibiofemoral OA grade 2 or higher, unilateral or bilateral
* Demonstrated knee OA related dysfunction per WOMAC score
* Not engaged in a regular exercise program for minimum of 6 months

Exclusion Criteria:

* Inability to obtain physician release for exercise
* High risk health status:

  e.g., uncontrolled medical conditions such as hypertension, diabetes, heart disease, pulmonary disease, high cholesterol, anginal type pain, dizziness or syncope, orthopnea or paroxysmal nocturnal dyspnea, ankle edema, heart palpitations or tachycardia, intermittent claudication, known heart murmur, unusual fatigue or shortness of breath with usual activities.
* Unresolved balance disorder
* Unresolved neurological disorder
* History of knee surgery or major knee trauma injury
* Hip or ankle instability, excessive weakness, surgery or major trauma injury
* Intra-articular joint injection within 4 weeks of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
WOMAC Osteoarthritis Scale; Function subscale change pre to post intervention - KBA vs. standard strength training | 8 weeks

SECONDARY OUTCOMES:
WOMAC subscale change in Pain and in Stiffness pre to post intervention | 8 weeks
Walking speed change in a timed Get Up & Go Test pre to post intervention | 8 weeks
Stair climbing and descending speed change pre to post intervention | 8 weeks
Gait quality measures with the GAITRite walking mat and EMG, pre to post intervention | 8 weeks
Spontaneous engagement in physical activity - change pre to post intervention as measured by the Human Activity Profile | 8 weeks
Efficacy for exercise change pre to post intervention as measured by the Self-Efficacy for Exercise scale. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Rogers, MS, Principal Investigator — The Arthritis Research Institute of America; Nauris Tamulevicius, PhD, Study Director — Morton Plant Mease Cheek-Powell Wellness Center; Frances V Wilder, PhD, Study Chair — The Arthritis Research Institute of America
Locations (1):
- Morton Plant Mease Cheek-Powell Wellness Center, Clearwater, Florida, United States